CLINICAL TRIAL: NCT06726590
Title: The Texas Interprofessional Pharmacogenomics Registry and Repository
Brief Title: Interprofessional Pharmacogenomics (IPGx) Registry and Repository
Acronym: IPGx Registry
Status: Recruiting | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY2023-0042
Record Dates: First submitted 2024-11-18; First posted 2024-12-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Cholesterol; Cancer; Blood Pressure Disorders; Heart Disease; Respiratory Ilness; COPD; Adverse Drug Reaction (ADR); Poly Pharmacy
Keywords: REGISTRY; REPOSITORY; POLYPHARMACY; ADVERSE DRUG REACTION
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms; Heart Diseases; Pulmonary Disease, Chronic Obstructive; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — blood, urine, and cheek cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Polypharmacy: Patients taking many medications or medications with severe side effects

SUMMARY:
This program collects genetic and health information to help doctors choose the right medications for patients.

DETAILED DESCRIPTION:
This study wants to understand how genes can affect how the body responds to medicines. This information will help us determine whether changing your medicine can make you healthier and improve your life. We will study your medical history for the last year and the next five years after you join the study.

study goals include:

* Enrolling patients who take multiple medications or have harmful side effects from their medications.
* Keeping all medical information and genetic samples from patients in one place.
* Helping doctors make better decisions about which medicines to prescribe.
* Influencing insurance companies and the government to help pay for this kind of medical care for people who need to change their medicine to stay healthy.

ELIGIBILITY:
Inclusion Criteria:

* The study will invite patients who are eligible for PGX workup/PGX care to participate, provided they meet the following criteria: Use of five or more medications, including over the counter drugs, supplements, natural products, cannabis products, or other recreational drugs, or
* Individuals taking blood pressure or depression medications, even if less than five medications.
* Ability to understand and give consent.
* Able to consent to donate blood and/or urine samples and buccal swabs.
* Able to answer detailed questionnaires, including quarterly questionnaires about ADRs, cognitive testing such as serial mini-mental status exams, and or quality of life questions.
* Able to understand that their health record and changes in health status will be followed for a five-year period and shared in deidentified form with the research community.
* All genders.
* Any age over 18 years.

Exclusion Criteria:

* Individuals admitted to hospice.
* Declines to participate or interact with staff/share their medical status.
* A diagnosis of Alzheimer's disease or related dementias in a medical record as this indicates a progressive, debilitating condition that impairs memory, thought processes, and functioning.,
* Individuals who are unable or unwilling to provide consent.
* Unable to verbally communicate and comprehend English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Texas A&M Health clinical programs.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and nature of ADRs on the Naranjo Scale | 5 years
  Patients will be referred to the Texas A&M Interprofessional Pharmacogenomics Clinic (IPGx) by their primary care physicians. A physician or ambulatory pharmacist in the IPGx clinic or Family Care Clinic will obtain a complete medical history, physical examination, and validate the patient's current concomitant medication list at the IPGx during the office visit. Patient medical information would be input into the CSN, which functions as a computable EHR medical record analysis, evaluation of polypharmacy status, and monitoring of Adverse Drug Reactions using the Naranjo Scale questionnaire will be conducted for the duration of the study.

SECONDARY OUTCOMES:
Serum/plasma drug concentrations | 5 years
  Patients will be referred to the Texas A&M Interprofessional Pharmacogenomics Clinic (IPGx) by their primary care physicians for an evaluation of pharmacokinetic and pharmacodynamic (PK/PD) assessments. For drug level measurement, urine samples will be collected using provided kits and shipped to the contracted laboratory via FedEx in biosafety shipping containers.

OTHER OUTCOMES:
Pharmacogenomic genotype with corresponding ADR phenotype | 5 years
  Patients will be referred to the Texas A&M Interprofessional Pharmacogenomics Clinic (IPGx) by their primary care physicians to evaluate genotyping and ADR. Clinical staff will obtain a buccal swab to collect DNA for a pharmacogenomic evaluation pursuant to the sample collection kits from the CLIA lab, which will occur at the start of the study period.
Drug-drug interactions, drug gene interactions, drug-drug-gene interactions | 5 years
  An assessment at the IPGx begins with a consultation by a pharmacist or physician. They will evaluate the medications and other drugs the patient is currently using, identifying any potential issues related to toxicity, drug interactions, or side effects that may be relevant to the patient's clinical presentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M Family Care, Bryan, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD deidentified